CLINICAL TRIAL: NCT05773313
Title: Social and Relational Capital to Overcome Social Determinants of Health.
Brief Title: A Study of Overcoming Social Determinants of Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Nathan L. Delafield, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22-012939; UL1TR002377 (NIH)
Record Dates: First submitted 2023-03-10; First posted 2023-03-17 (Actual); Results first posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Social Determinants of Health (SDOH)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The Open Table Model (Experimental): Subjects identified as having their health negatively impacted by Social Determinants of Health (SDOH) will meet with The Open Table members to determine their specific needs, decide on a plan for overcoming this need and following up to ensure resolution.
  Interventions: Behavioral: The Open Table

INTERVENTIONS:
Behavioral: The Open Table — An organization that connects community volunteers to individuals in need to help overcome life's challenges.

SUMMARY:
This study is being done to determine if assistance in accessing community resources can improve health outcomes. Social determinants of health are the conditions in which individuals are born, work and live that can impact health. These can include access to healthcare, healthy food, education, safe neighborhoods, transportation, political and social environments that are safe and fair.

ELIGIBILITY:
Inclusion Criteria:

- Identified social determinants of health (SDOH). need that impacts healthcare outcomes (identified by the healthcare team)

Exclusion Criteria:

* Non-english speaking patients
* Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Delafield, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- The Open Table Model: Subjects identified as having their health negatively impacted by Social Determinants of Health (SDOH) met with The Open Table members to determine their specific needs, decide on a plan for overcoming this need and following up to ensure resolution.
  The Open Table: An organization that connects community volunteers to individuals in need to help overcome life's challenges.
Period: Overall Study
Arm/Group | The Open Table Model
Started | 12
Completed | 9
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | The Open Table Model
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (18.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 7
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Participant Center for Medicare and Medicaid Services (CMS) Accountable Health Social Determinants of Health (SDOH) Screening Assessment
Description: Evaluated using the CMS Accountable Health SDOH Screening Tool used to assess patient needs across the following domains: house instability, food insecurity, transportation problems, utility help needs, interpersonal safety, financial strain, employment, family and community support, education, physical activity, substance use, mental health, and disabilities that community services can help with. If the participant chose the underlined option, they might have an unmet health-related social need. Only domains where an unmet health-related social need was identified was included in the analysis.
Time Frame: Baseline and 12 months
Population: 3 participants did not complete the CMS accountable health SDOH screening assessment at 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | The Open Table Model
Number analyzed (Participants) | 12
Participants
  Food Insecurity-Baseline | 6
  Food Insecurity-12 Months: number analyzed (Participants) | 9
  Food Insecurity-12 Months | 5
  Financial Strain-Baseline | 9
  Financial Strain-12 Months: number analyzed (Participants) | 9
  Financial Strain-12 Months | 5
  Family and Community Support-Baseline | 10
  Family and Community Support-12 Months: number analyzed (Participants) | 9
  Family and Community Support-12 Months | 7
  Physical Activity-Baseline | 9
  Physical Activity-12 Months: number analyzed (Participants) | 9
  Physical Activity-12 Months | 7
  Disability-Baseline | 12
  Disability-12 Months: number analyzed (Participants) | 9
  Disability-12 Months | 8
Statistical Analysis 1: Comparison: The Open Table Model; Food Insecurity; Test type: Superiority; p > 0.999, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: The Open Table Model; Financial Insecurity; Test type: Superiority; p = 0.250, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: The Open Table Model; Social Isolation; Test type: Superiority; p > 0.999, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: The Open Table Model; Physical Inactivity; Test type: Superiority; p > 0.999, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: The Open Table Model; Disability; Test type: Superiority; p > 0.999, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Change in Resilience
Description: Evaluated using the 6-item Brief Resilience Scale (BRS) questionnaire assessing the participants ability to bounce back on a 1-5 scale range. Total questions scores are divided by total number of questions answered for a final score range from 1.00-2.99 = low resilience; 3.00-4.30 = normal resilience; 4.31-5.00 = high resilience.
Time Frame: Baseline and 12 months
Population: 3 participants did not complete the BRS questionnaire at 12 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Open Table Model
Number analyzed (Participants) | 12
score on a scale
  Baseline | 3.0 (0.94)
  12 Months: number analyzed (Participants) | 9
  12 Months | 3.3 (0.98)
Statistical Analysis 1: Comparison: The Open Table Model; Test type: Superiority; p = 0.461, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Hospitalizations
Description: Difference in total number of hospitalizations in the 12 months before intervention and 12 months during intervention.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: Hospitalizations
Arm/Group | The Open Table Model
Number analyzed (Participants) | 12
Hospitalizations
  Baseline | 0.3 (0.62)
  12 Months | 0.3 (0.89)
Statistical Analysis 1: Comparison: The Open Table Model; Test type: Superiority; p > 0.999, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Emergency Room Visits
Description: Difference in total number of emergency room visits in the 12 months before intervention and 12 months during intervention.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: Visits
Arm/Group | The Open Table Model
Number analyzed (Participants) | 12
Visits
  Baseline | 1.7 (1.50)
  12 Months | 1.2 (1.85)
Statistical Analysis 1: Comparison: The Open Table Model; Test type: Superiority; p = 0.438, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Primary Care Visits
Description: Difference in total number of primary care visits in the 12 months before intervention and 12 months during intervention.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: Visits
Arm/Group | The Open Table Model
Number analyzed (Participants) | 12
Visits
  Baseline | 8.3 (6.94)
  12 Months | 5.5 (5.32)
Statistical Analysis 1: Comparison: The Open Table Model; Test type: Superiority; p = 0.080, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time of informed consent through study completion, approximately 12 months.
Description: Only adverse events related to the intervention were collected.
Arm/Group | The Open Table Model
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT05773313/Prot_SAP_000.pdf